CLINICAL TRIAL: NCT03003546
Title: LS1681: A Phase I Trial of AR160 (Abraxane/Rituximab 160nm Nanoparticle) in Relapsed/Refractory B Cell Lymphomas Including Transformed Follicular Lymphoma
Brief Title: Nab-paclitaxel/Rituximab-coated Nanoparticle AR160 in Treating Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma, LS1681 Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS1681; NCI-2016-01984 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA097274 (NIH)
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Aggressive Non-Hodgkin Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Aggressive Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 130-nm albumin-bound paclitaxel; Rituximab; Nanoparticles; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (AR160) (Experimental): Patients receive nab-paclitaxel/rituximab-coated nanoparticle AR160 IV over 30-60 minutes on days 1, 8, and 15. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nab-paclitaxel/Rituximab-coated Nanoparticle AR160; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab-paclitaxel/Rituximab-coated Nanoparticle AR160 — Given IV
  Other Names: Abraxane coated with Rituximab; Abraxane Coated with Rituximab 160nm Nanoparticle; Abraxane/Rituxan 160 Complex; AR160
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the best dose and side effects of paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel)/rituximab-coated nanoparticle AR160 in treating patients with B-cell non-Hodgkin lymphoma that has come back (relapsed) or is not responding to treatment (refractory). Nab-paclitaxel/rituximab-coated nanoparticle AR160 is a combination of paclitaxel albumin-stabilized nanoparticle formulation and rituximab. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with rituximab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving paclitaxel albumin-stabilized nanoparticle formulation and rituximab may work better in treating patients with B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the maximum tolerated dose (MTD) of nab-paclitaxel/rituximab-coated nanoparticle AR160 (AR160) in patients with relapsed/refractory B-cell non-Hodgkin lymphoma (NHL). (Phase I)

SECONDARY OBJECTIVES:

I. To assess the toxicity and safety of AR160. II. To assess complete response rate (CR) progression free survival (PFS), and overall survival (OS) of AR160 with relapsed/refractory B-cell NHL.

CORRELATIVE RESEARCH OBJECTIVE:

I. Evaluate pharmacokinetics (PK) of AR160 in two formal PK studies, dose 1 of cycle 1 (48 hours [h] PK analysis) and dose 1 of cycle 2 (24h PK analysis). As of Amendment 4, PKs will no longer be collected.

OUTLINE: This is a dose-escalation study.

Patients receive nab-paclitaxel/rituximab-coated nanoparticle AR160 intravenously (IV) over 30-60 minutes on days 1, 8, and 15. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Histological confirmation of relapsed/refractory B-cell NHL, CD20+

  * NOTE: patients with small lymphocytic lymphoma (SLL) are eligible however patients with chronic lymphocytic leukemia (CLL) are not eligible
  * Waldenstrom macroglobulinemia patients are not eligible; aggressive lymphoma patients who are transplant eligible must have undergone a transplant
  * The biopsy confirming relapse can be up to 24 weeks prior to registration as long as there is no intervening therapy
* Measurable disease (at least 1 lesion of >= 1.5 cm in one diameter) as detected by computed tomography (CT) or the CT images of the positron emission tomography (PET)/CT. Skins lesions can be used if the area is greater than or equal to 2 cm in at least one diameter and photographed with a ruler
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 14 days prior to registration)
* Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) or if total bilirubin is > 1.5 X ULN, the direct bilirubin =< ULN (obtained =< 14 days prior to registration)
* Alkaline phosphatase =< 3 X ULN unless due to direct lymphoma involvement, and then =< 5 X ULN (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST) =< 3 X ULN unless due to direct lymphoma involvement, and then =< 5 X ULN (obtained =< 14 days prior to registration)
* Calculated creatinine clearance must be >= 30 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Life expectancy >= 3 months
* Ability to provide written informed consent
* Willing to return to enrolling institution for follow-up (during the treatment phase of the study)
* Willing to provide blood samples for correlative research purposes
* Failed or are intolerant to 2 or more lines of established therapy or for whom no other treatment options are available in the opinion of the investigator
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Disease-free of prior invasive malignancies for > 5 years prior to registration

  * Note: Exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Active central nervous system (CNS) lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells that requires therapy
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Received most recent therapy =< 4 weeks prior to registration; NOTE: use of systemic steroid therapy is allowed pretreatment
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Patients with >= 25% of the bone marrow radiated for other diseases
* Other medical conditions including but not limited to:

  * History of liver disease such as cirrhosis, chronic active hepatitis, chronic persistent hepatitis or hepatitis B or C
  * Active infection requiring parenteral antibiotics
  * New York Heart Association class II-IV congestive heart failure (serious cardiac arrhythmia requiring medication)
  * Myocardial infarction or unstable angina =< 6 months prior to registration
  * Congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
  * Clinically significant peripheral vascular disease
  * History of CNS disease (e.g., primary brain tumor, vascular abnormalities, etc.), clinically significant stroke or transient ischemic attack (TIA) =< 6 months prior to registration, seizures not controlled with standard medical therapy
  * Neuropathy ˃ grade 3
* Administration of strong CYP2C8 or CYP3A4 inhibitors or inducers =< 10 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 28 days
  MTD will be defined as the highest dose level patients develop a dose limiting toxicity assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The maximum grade of each type of toxicity will be recorded for each patient. For each toxicity reported by dose level, the percentage of patients developing any degree of that toxicity as well as the percentage of patients developing a severe degree (grade 3 or higher) will be determined.

SECONDARY OUTCOMES:
Tumor response | Up to 2 years
  Will be assessed using the Lugano Classification Response criteria. A table will be constructed to display by dose level, the number of patients treated at that dose level, the number of cycles of treatment administered, dose limiting toxicity (DLT) observed, and number of responses.
Progression free survival | Time from registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 2 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Overall survival | Time from registration to death due to any cause, assessed up to 2 years
  The distribution of overall survival will be estimated using the method of Kaplan Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Habermann, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials